CLINICAL TRIAL: NCT03862443
Title: Influence of Financial Incentives on Oral Disease Management in Young Children: A Randomized Pilot Trial
Brief Title: BEhavioral EConomics for Oral Health iNnovation Pilot Trial
Acronym: BEECON Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-19968
Record Dates: First submitted 2019-02-14; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Toothbrushing; Dental Plaque; Parent-Child Relations; Oral Hygiene; Dental Caries
Keywords: Preventive Dentistry; Health Disparities; Health Behavior; Behavioral Economics; Monetary Incentives
MeSH Terms: conditions — Dental Plaque; Dental Caries; Health Behavior

STUDY DESIGN:
Intervention Model Description: Eligible consenting parent-child participant dyads, within strata and permuted blocks, will be randomized in equal allocation to one of three arms. Strata will be based on smartphone operating system (iOS or Android).
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent outcomes assessor and PIs will be blinded to participants' group assignment, and participants will be told that the examiner and PIs cannot answer any incentive questions and they should not mention the incentive program to them. (Due to the nature of the intervention, the staff explaining the study arms after randomization and providing the incentive gift cards at follow-up visits cannot be blinded.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fixed Incentive (Experimental): Eligible to earn a weekly payment during the 2-month incentive intervention period. Possible weekly winnings depend on toothbrushing performance collected through smart powered toothbrush synced to a smartphone app: low adherence threshold (brushing child's teeth once per day for 7 days in a week) will win $5; high adherence threshold (brushing twice per day for 14 days in a week) will win $10.
  Interventions: Behavioral: Fixed Incentive
- Drawing Incentive (Experimental): Eligible to earn a weekly drawing entry with different winning probabilities during the 2-month incentive intervention period. Possible weekly winnings depend on toothbrushing performance collected through smart powered toothbrush synced to a smartphone app: low adherence threshold (brushing child's teeth once per day for 7 days in a week) will have an 18% chance of winning $25 and a 1% chance of winning $50 (expected $5 payout); high adherence threshold (brushing twice per day for 14 days in a week) will have a 34% chance of winning $25 and a 3% chance of winning $50 (expected $10 payout).
  Interventions: Behavioral: Drawing Incentive
- Control - Delayed Incentive (No Intervention): No rewards during the first 2-months, but information on toothbrushing performance collected through smart powered toothbrush synced to a smartphone app. After the Month 2 follow-up visit, may opt to participate in a delayed 2-month open label extension to earn the same monetary rewards the fixed incentive intervention group could earn Baseline through Month 2. Not a formal part of this trial, but rather a necessary condition to assure all participating parents/caregivers have the chance to earn the same monetary incentives.

INTERVENTIONS:
Behavioral: Fixed Incentive — The Fixed Incentive intervention is a fixed reward, in which participants are eligible for fixed weekly payments based on toothbrushing performance collected through smart powered toothbrush synced to a smartphone app.
  Arms: Fixed Incentive
Behavioral: Drawing Incentive — The Drawing Incentive intervention is a drawing reward, in which participants are eligible for weekly payments based on toothbrushing performance collected through smart powered toothbrush synced to a smartphone app.
  Arms: Drawing Incentive

SUMMARY:
This Phase I randomized pilot trial will assess the efficacy of a fixed incentive payment program and drawing incentive payment program versus a control program to promote early childhood caries (ECC) preventive health behaviors (i.e., toothbrushing performance and dental visit attendance) for young children of predominantly Latino parents/caregivers enrolled in/waitlisted for Early Head Start (EHS) home visit programs.

DETAILED DESCRIPTION:
If both groups are acceptable and feasible, the reward group with toothbrushing outcomes at least 20% better than the other one (and the control) will be chosen for a future Phase II/III trial; if they are similar, the fixed monetary reward will be used because it is simpler to explain, monitor, and implement.

ELIGIBILITY:
Inclusion Criteria for Parent/Caregiver:

* Provide signed and dated informed consent form in English or Spanish.
* Agree to comply with all study procedures and be available for the duration of the study visit.
* Male or female, aged 18 and older.
* Speak, read, and write either English or Spanish.
* Be a parent or caregiver of a child at least 6 months old but less than 3.5 years (42 months), with at least 2 fully erupted teeth and enrolled in, or waitlisted for, one of the three participating Los Angeles County EHS home visit programs.
* Not be planning to move residence for the next 6 months outside the greater Los Angeles area.
* Own a smartphone with the Google Play or iTunes store and be willing to download the smart powered TB app
* Be willing to be contacted via text-messaging (SMS) for study related notifications, such as incentives earned or reminders to sync the TB

Exclusion Criteria:

* Known allergic reaction to components of the study product(s).
* Uncooperative or behaviorally unsuited (assessed during a TB prophylaxis at the initial baseline study visit).
* A sibling of a child already enrolled in the study (the family's oldest child in the eligible age range will be the study child).
* Enrolled in foster care.
* Anything else that would place him/her at increased health risk or preclude the individual's full compliance with or completion of the study.

Ages: 6 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-08-13 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Mean number of qualifying half-day toothbrushing episodes per week | Baseline visit through the Month 2 visit
  Mean number of qualifying half-day episodes per week in which a parent/caregiver brushes a child's teeth. (A Bluetooth-recorded toothbrushing episode qualifies if it lasts at least one minute within one of 14 half-day windows in the week.)
Proportion of parents/caregivers attending a dental visit | Month 2 visit
  In the subset of children at baseline with no dental visit in the EHS ChildPlus health module, whether or not the child has a ChildPlus documented dental visit at the two-month follow-up.

SECONDARY OUTCOMES:
Proportion of weeks the parent/caregiver synced toothbrushing data with the app | Baseline visit through Month 2 visit
  Proportion of weeks the parent/caregiver synced toothbrushing data with the app
Mean number of days per week with parent/caregiver-reported twice daily brushing | Baseline visit through the Month 2 visit
  Twice daily brushing with fluoridated toothpaste, based on parent/caregiver-reported frequency diaries
Fluoridated toothpaste use | Baseline visit through the Month 2 visit
  Change in child toothpaste pump weight
Child plaque score | Month 2 visit
  The child's Debris Index component (plaque score) of the Simplified Oral Hygiene Index (Greene and Vermillion) modified to include only maxillary incisor teeth after disclosing with plaque solution. The scale (which is a mean value) range is 0 (no debris or stain) to 3 (soft debris covering more than two thirds of the exposed tooth surface).
EHS site participation | Month 0
  Willingness of LA County EHS to sign memoranda of understanding
EHS staff participation | Month 0
  Willingness of EHS staff participation in assisting with recruitment
Proportion of parents/caregivers who consent | Baseline visit
  Willingness of parents/caregivers to provide informed consent and approve access to ChildPlus dental visit data
Proportion of parents/caregivers willing to be randomized | Baseline visit
  Willingness of parents/caregivers to be randomized to a study arm as part of the consenting process
Proportion of parents/caregivers adhering to study procedures | Baseline visit through the Month 2 visit
  Willingness of parents/caregivers to adhere to study procedures, including completing questionnaire instruments, bringing toothbrushing frequency diaries to 2-month follow-up visit, and bringing toothpaste pump to 2-month follow-up visit
Proportion of children who cooperate | Baseline visit through the Month 2 visit
  Willingness of child to cooperate with study procedures, including dental screening, extraoral photo, and plaque assessment
Proportion of parents/caregivers willing to use the toothpaste pump | Baseline visit through the Month 2 visit
  Willingness to use the toothpaste pump (percentage with any use and percentage change in pump weight)
Feasibility of measuring toothbrushing frequency with diaries | Month 2 visit
  Bringing toothbrushing diaries to the follow-up visit and willingness to provide them to study staff
Feasibility of using toothpaste pump weight as a measure of usage | Month 2 visit
  Bringing the toothpaste pump to the follow-up visit for weighing
Proportion of parents/caregivers willing to use the disclosing solution | Baseline visit and Month 2 visit
  Willingness of children to comply with the plaque disclosing procedure
Proportion of parents/caregivers willing to use photographs for central assessment | Baseline visit and Month 2 visit
  Willingness of the child to allow photographs, the ability to transmit the photographs securely, and the ability of the central clinician to score them reliably and confidently
Proportion of parents/caregivers willing to use smart powered toothbrush | Baseline visit through Month 2 visit
  Willingness to use the smart powered toothbrush handle (percentage with any brushing data)
Comfort with smart powered toothbrush | Baseline visit through Month 2 visit
  Child and parent comfort level with using the smart powered toothbrush
Proportion of parents/caregivers willing to use smartphone app | Baseline visit
  Willingness to download the smartphone app and keep it for the duration of the study
Proportion of parents/caregivers willing to receive text messages | Baseline visit
  Willingness to be contacted with study-related text messages each week during the intervention period
Feasibility of syncing toothbrush to app | Baseline visit
  Successfully synced the toothbrush to app during baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Gansky, DrPH, Principal Investigator — University of California, San Francisco; Francisco Ramos-Gomez, DDS, MS, MPH, Principal Investigator — University of California, Los Angeles; James G Kahn, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Venice Family Clinic Children First Early Head Start, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] White JS, Ramos-Gomez F, Liu JX, Jue B, Finlayson TL, Garza JR, Crawford AH, Helman S, Santo W, Cheng J, Kahn JG, Gansky SA. Monetary incentives for improving smartphone-measured oral hygiene behaviors in young children: A randomized pilot trial. PLoS One. 2020 Jul 30;15(7):e0236692. doi: 10.1371/journal.pone.0236692. eCollection 2020. PMID 32730310